CLINICAL TRIAL: NCT01510392
Title: Prospective Evaluation of Optical Coherence Tomography Usage in the Screening of Eye Diseases
Brief Title: CEI Van Outreach Screening Study
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, Michael Chiang, MD, Professor, Provisional, Department of Ophthalmology and Medical Informatics & Clinical Epidemiology, Oregon Health and Science University
Other Study IDs: OHSU IRB#00008034-Outreach
Record Dates: First submitted 2012-01-03; First posted 2012-01-16 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Glaucoma; Macular Disease; Keratoconus
Keywords: Optical coherence tomography; Glaucoma; Macula; Keratoconus; Screening
MeSH Terms: conditions — Glaucoma; Macular Degeneration; Keratoconus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: OCT imaging, the FDA Cleared iVue — The OCT system scans a beam of light across the eye to take a picture. OCT imaging does not touch the eye. This is a test that is performed using an FDA approved system, and is regularly used to take pictures of the back of the eye.

SUMMARY:
The primary goal of the trial is to show that optical coherence tomography (OCT) technology can be used to effectively screen for diseases of the eye including glaucoma, macular diseases and keratoconus. Glaucoma is a disease that causes permanent vision loss and is usually accompanied by increased eye pressure. Macular diseases affect sharp, central vision. Keratoconus is a disease that affects the cornea (clear surface covering the colored part of the eye).

DETAILED DESCRIPTION:
The identification of many eye diseases would significantly benefit from earlier detection than is available with typical eye exams. Optical coherence tomography (OCT) is an imaging technology that can perform non-contact cross-sectional imaging of tissue structure in real time. It is similar to ultrasound B-mode imaging, except that OCT measures the intensity of reflected light rather than sound waves.

ELIGIBILITY:
Inclusion Criteria:

* Participant undergoing a screening examination at the Casey Eye Institute Outreach Van.
* Participants must be between the ages of 18 and 89 years old.

Exclusion Criteria:

* Inability to give informed consent.
* Inability to maintain stable fixation for OCT imaging

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be performed enrolling participants from the Casey Eye Institute outreach van.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2012-01; Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
OCT screening efficacy for detection of early stage eye diseases in comparison to the current standard of care methods | 1 year
  The primary goal of the trial is to show that OCT technology, specifically the FDA cleared iVue, can be used to effectively screen for glaucoma, macular diseases and keratoconus. The rate of detection of these diseases detected using OCT will be compared to the rate of detection by the physician's exam.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chiang, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Casey Eye Institute Outreach Screening Van, Portland, Oregon, United States